CLINICAL TRIAL: NCT02393599
Title: Phase 1, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess Potential Interactions Between Intravenous Cocaine and Oral Lorcaserin
Brief Title: Study to Assess Potential Interactions Between Intravenous Cocaine and Oral Lorcaserin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Lorcaserin-Phase 1b-001
Record Dates: First submitted 2015-03-04; First posted 2015-03-19 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2015-10

CONDITIONS: Cocaine Abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lorcaserin (Experimental): Lorcaserin (10mg) will be administered 2 times per day from Days 3 to 9 and only one time on Day 10
  Interventions: Drug: Lorcaserin; Drug: Cocaine Infusion
- Placebo (Placebo Comparator): Placebo will be administered 2 times per day from Days 3 to 9 and only one time on Day 10
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorcaserin — 10 mg 2 times per day from Day 3 to 9 and one time on Day 10
  Arms: Lorcaserin
Drug: Placebo — 10 mg 2 times per day from Day 3 to 9 and one time on Day 10
  Arms: Placebo
Drug: Cocaine Infusion — Screening / Session 1, Study Day -2: 20 mg cocaine, followed by a saline infusion, followed by 40 mg cocaine Baseline/ Session 2, Study Day 1: Saline or 20 mg cocaine followed by either 20 mg cocaine or saline Baseline / Session 3, Study Day 2: Saline or 40 mg cocaine followed by either 40 mg cocaine or saline Treatment / Session 4, Study Day 9: Saline or 20 mg cocaine followed by either 20 mg cocaine or saline Treatment / Session 5, Study Day10: Saline or 40 mg cocaine followed by either 40 mg cocaine or saline
  Arms: Lorcaserin

SUMMARY:
The primary objective of this study is to determine if there are significant interactions between oral lorcaserin treatment concurrent with 20 and 40 mg intravenous (i.v.) cocaine infusions by measuring adverse events (AEs) and cardiovascular responses including heart rate (HR), blood pressure (BP), and electrocardiogram (ECG) (including QTc).

ELIGIBILITY:
Inclusion Criteria:

* Be volunteers who are not seeking treatment for drug addiction.
* Be between 18 and 50 years-of-age.
* Meet Diagnostic and Statistical Manual (DSM-IV) - Text Revision (TR) criteria for current cocaine abuse as assessed using the MINI neuropsychiatric interview (version 6.0).
* Have a body mass index (BMI) within a range of 18.0 to 34.0 kg/m2 and a minimum weight of at least 50.0 kg at screening.
* Have experience using cocaine by the smoked or i.v. route at least 6 times in the past 12 months prior to clinic intake (Day -3) and at least one use within the past 30 days.
* Provide a urine sample positive for cocaine at least once during screening (Days -28 to -4).
* Be able to verbalize understanding of consent form, able to provide written informed consent, and verbalize willingness to complete study procedures.
* Females must have a negative serum pregnancy test at screening and negative urine pregnancy test at intake prior to receiving the first dose of investigational drug. They must also be postmenopausal, have had a hysterectomy, been sterilized, have a partner with a vasectomy, or agree to use one of the following methods of birth control starting at least 14 days prior to clinic intake:

  1. diaphragm and condom by partner
  2. condom and spermicide by partner
  3. intrauterine device and condom by partner
  4. sponge and condom by partner
  5. complete abstinence from sexual intercourse
  6. oral contraceptives, Depo-Provera, Norplant, Patch, and intrauterine progesterone contraceptive
* Be able to comply with protocol requirements, rules and regulations of the study site and be likely to complete all the study treatments.

Exclusion Criteria:

* Please contact site directly for more information

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | From intake (day -3) through follow-up (day 26)
Number of Participants with Cardiovascular Responses | From screening (day -28 through day -4) through follow-up (day 26)

SECONDARY OUTCOMES:
Number of Participants with an Change in the Pharmacokinetics (PK) of Cocaine by Measuring the Cocaine Concentration in Plasma | Day 4, 6, 8 through 12

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, Ph.D., Principal Investigator — Vince & Associates Clinical Research, Inc.
Locations (1):
- Vince Associates Clinical Research, Inc., Overland Park, Kansas, United States